CLINICAL TRIAL: NCT00773734
Title: A Phase 2B, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Efficacy and Safety Study of Apremilast (CC-10004) in Subjects With Moderate-to-Severe Plaque-Type Psoriasis (Core Study)
Brief Title: Efficacy and Safety Study of Apremilast (CC-10004) in Subjects With Moderate-to-Severe Plaque-Type Psoriasis (Core Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-005; NCT00953875 (obsolete NCT alias); NCT01130116 (obsolete NCT alias)
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis; Plaque-type Psoriasis
Keywords: moderate-to-severe plaque-type psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Apremilast 10mg (Experimental): Apremilast 10 mg administered orally twice daily (BID) for 16 weeks (following dose titration) during the placebo controlled phase followed by 10 mg Apremilast tablets orally administered BID for 8 weeks in the active treatment phase
  Interventions: Drug: Apremilast 10mg
- Apremilast 20mg (Experimental): Apremilast 20 mg administered orally twice daily (BID) for 16 weeks (following dose titration) during the placebo controlled phase followed by 20 mg Apremilast tablets orally administered BID for 8 weeks in the active treatment phase
  Interventions: Drug: Apremilast 20mg
- Apremilast 30 mg (Experimental): Apremilast 30 mg administered orally twice daily (BID) for 16 weeks (following dose titration) during the placebo controlled phase followed by 30 mg Apremilast tablets orally administered BID for 8 weeks in the active treatment phase
  Interventions: Drug: Apremilast 30 mg
- Placebo (Placebo Comparator): Oral Placebo tablets administered twice daily (BID) for 16 weeks during the placebo-controlled phase.
  Interventions: Drug: Placebo
- Placebo/Apremilast 20 mg (Experimental): Participants initially randomized to receive placebo twice daily during the 16 week placebo controlled phase are re-randomized to 20 mg apremilast BID during the 8 week active treatment phase
  Interventions: Drug: Apremilast 20mg
- Placebo/Apremilast 30mg (Experimental): Participants initially randomized to receive placebo twice daily during the 16 week placebo controlled phase are re-randomized to 30 mg apremilast BID during the 8 week active treatment phase
  Interventions: Drug: Apremilast 30mg

INTERVENTIONS:
Drug: Apremilast 10mg
  Other Names: Apremilast tablets; CC-10004; Otezla
  Arms: Apremilast 10mg
Drug: Apremilast 20mg
  Other Names: Apremilast tablets; CC-10004; Otezla
  Arms: Apremilast 20mg
Drug: Apremilast 30 mg
  Other Names: Apremilast tablets; CC-10004; Otezla
  Arms: Apremilast 30 mg
Drug: Placebo
  Arms: Placebo
Drug: Apremilast 30mg
  Other Names: Apremilast tablets; CC-10004; Otezla
  Arms: Placebo/Apremilast 30mg
Drug: Apremilast 20mg
  Other Names: Apremilast tablets; CC-10004; Otezla
  Arms: Placebo/Apremilast 20 mg

SUMMARY:
The purpose of this study was to test if the drug apremilast was safe, if it helped improve psoriasis, and how well the participants tolerated it.

DETAILED DESCRIPTION:
This study fully explored the extent of treatment benefit achieved with doses of apremilast up to 30 mg by mouth (PO) twice daily (BID) with treatment duration for up to 6 months. In addition, it was important to determine the minimally effective dose for apremilast and more fully elucidate the dose response curve in this patient population. The results from this study helped guide the selection of the dose in the phase 3 trials.

Participants meeting eligibility criteria at the Baseline Visit (Week 0) were centrally randomized with the use of a permuted-block randomization list, with equal allocation to each of the four treatment arms: 10 mg, 20 mg or 30 mg PO BID of apremilast or placebo. In an effort to mitigate the dose-dependent adverse effects of apremilast (e.g., headache or gastrointestinal disturbances), participants had their dose titrated over a 7-day period (Days 1 through7). Participants received 10 mg PO BID of apremilast or identically-appearing placebo during Days 1 to 2. Participants randomized to the 10 mg BID dose continued taking this dose throughout the treatment phase of the study. Those participants randomized to the 20 mg BID dose were dose titrated to 20 mg PO BID of apremilast or identically-appearing placebo during Days 3 to 4 of dosing. Participants randomized to the 20 mg BID dose continued taking this dose throughout the treatment phase of the study. Those participants randomized to the 30 mg BID dose were dose titrated to 30 mg PO BID of apremilast or identically-appearing placebo during Days 5 to 7 and continued taking this dose throughout the treatment phase of the study. At Week 16, all participants originally randomized to the placebo arm were re-randomized to 20 mg BID or 30 mg BID of apremilast. All participants (i.e., those that were continuing their Apremilast dosing regimen, as well as those that were switched from placebo to apremilast) received drug at Week 16 in a treatment arm in a blinded fashion. In addition, participants who transitioned from placebo to active medication at Week 16 completed a dose titration schedule to help mitigate any potential GI side effects that may have jeopardized the blinding of the treatment arms.

At Week 24 (end of core study and beginning of an extension study), participants were given the option to enroll into an extension study (PSOR-005E NCT00953875) and continue on the same apremilast dosage they had received at the end of the core study, during Weeks 24-52, a total of 28 weeks. Participants who elected not to enter into the treatment extension study, completed a 4-week observational follow-up phase of the core study. At Week 52 (end of extension study and beginning of a long-term extension study), participants were given the option to enroll into a long term extension study (PSOR-005LTE NCT01130116), for 4 additional years. Participants who were treated with apremilast 10 mg BID in the extension study were randomly assigned and dose titrated to either apremilast 20 mg BID or 30 mg BID. Participants who were dosed with 20mg or 30 mg BID in the extension study continued to receive the same dose in the long-term extension study. The long-term extension study is anticipated to complete in May 2016.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* ≥18 years of age at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements.
* Diagnosis of chronic, stable plaque psoriasis at least 6 months prior to screening as defined by:

  1. PASI (Psoriasis Area and Severity Index) score ≥ 12
  2. Body Surface Area (BSA) ≥ 10%
* Candidate for photo/systemic therapy
* In good health as judged by the investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), serum chemistry, hematology, immunology, and urinalysis
* Meet all laboratory criteria as defined per protocol
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening (Visit 1). In addition, sexually active FCBP must agree to use TWO of the following adequate forms of contraception methods. A FCBP must agree to have pregnancy tests every 4 weeks while on study medication
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with FCBP while on study medication and for 84 days after taking the last dose of study medication

Exclusion Criteria:

* History of clinically significant disease (as determined by the investigator)
* Pregnant or breastfeeding
* History of active mycobacterial infection within 3 years
* History of Human Immunodeficiency Virus (HIV) infection
* Congenital and acquired immunodeficiencies
* Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening
* Antibodies to Hepatitis C at screening
* Malignancy or history of malignancy except for treated [i.e., cured] basal-cell skin carcinomas
* Any condition, including the presence of laboratory abnormalities, that places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Psoriasis flare within 4 weeks of screening
* Topical therapy within 2 weeks of randomization
* Systemic therapy for psoriasis within 4 weeks of randomization
* Use of phototherapy within 4 weeks of randomization [(i.e., Ultraviolet (UVB), Psoralens and long-wave ultraviolet radiation (PUVA)]
* Adalimumab, etanercept, efalizumab or infliximab within 12 weeks of randomization
* Alefacept within 24 weeks of randomization
* Investigational drug within 4 weeks of randomization, or 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer)
* Prolonged sun exposure or use of tanning booths or other ultraviolet light sources

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2009-08-01 (Actual); Study Completion 2015-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (35):
- United States (20):
  - Associates In Research Inc, Fresno, California
  - Dermatology Associates, Los Angeles, California
  - Stanford University School of Medicine, Redwood City, California
  - Atlantic Skin & Cosmetic Surgery Group, PC, Wilmington, Delaware
  - Renstar Medical Research, Ocala, Florida
  - Atlanta Dermatology, Vein & Research Center, Alpharetta, Georgia
  - NorthShore University HealthSystem, Skokie, Illinois
  - Dawes/Fretzin Dermatology Group Inc, Indianapolis, Indiana
  - Dermatology & Advanced Aesthetics, Lake Charles, Louisiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Central Dermatology, St Louis, Missouri
  - UMDNJ Robert Wood Johnson, New Brunswick, New Jersey
  - Wright State University, Dayton, Ohio
  - Allergy, Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - Northwest Cutaneous Research Specialists, Portland, Oregon
  - Oregon Med. Research Center, PC, Portland, Oregon
  - Rivergate Dermatology Clinical Research, Goodlettsville, Tennessee
  - Modern Research Associates, Dallas, Texas
  - Dermatology Associates of Seattle, Seattle, Washington
  - Aurora Advanced Healthcare, Inc, Milwaukee, Wisconsin
- Canada (15):
  - Stratica Medical, Edmonton, Alberta
  - Dr. Lorne E. Albrecht, Surrey, British Columbia
  - Alpha Clinical Research Centre, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Associates, Halifax, Nova Scotia
  - Ultranova Skincare, Barrie, Ontario
  - Dermatrials Research Division, Hamilton, Ontario
  - Guenther Dermatology Research Centre, London, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Dr. Michael Robern, Ottawa, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - XLR8 Research, Windsor, Ontario
  - Innovaderm Research Laval Inc., Laval, Quebec
  - Centre De Recherche Dermatologique du Qu, MetSte-Foy, Quebec
  - Innovaderm Research Inc., Montreal, Quebec
  - International Dermatology Research, Inc., Montreal, Quebec

REFERENCES:
- [Background] Papp K, Cather JC, Rosoph L, Sofen H, Langley RG, Matheson RT, Hu C, Day RM. Efficacy of apremilast in the treatment of moderate to severe psoriasis: a randomised controlled trial. Lancet. 2012 Aug 25;380(9843):738-46. doi: 10.1016/S0140-6736(12)60642-4. Epub 2012 Jun 29. PMID 22748702
- [Background] Ohtsuki M, Kubo H, Morishima H, Goto R, Zheng R, Nakagawa H. Guselkumab, an anti-interleukin-23 monoclonal antibody, for the treatment of moderate to severe plaque-type psoriasis in Japanese patients: Efficacy and safety results from a phase 3, randomized, double-blind, placebo-controlled study. J Dermatol. 2018 Sep;45(9):1053-1062. doi: 10.1111/1346-8138.14504. Epub 2018 Jun 15. PMID 29905383
- [Background] Knuckles MLF, Levi E, Soung J. Defining and treating moderate plaque psoriasis: a dermatologist survey. J Dermatolog Treat. 2018 Nov;29(7):658-663. doi: 10.1080/09546634.2018.1443200. Epub 2018 Mar 22. PMID 29502473
- [Background] Knuckles MLF, Levi E, Soung J. Treating moderate plaque psoriasis: prospective 6-month chart review of patients treated with apremilast. J Dermatolog Treat. 2019 Aug;30(5):430-434. doi: 10.1080/09546634.2018.1528326. Epub 2018 Nov 26. PMID 30339049
- [Background] Wu JJ, Pelletier C, Ung B, Tian M. Real-world treatment patterns and healthcare costs among biologic-naive patients initiating apremilast or biologics for the treatment of psoriasis. J Med Econ. 2019 Apr;22(4):365-371. doi: 10.1080/13696998.2019.1571500. Epub 2019 Feb 4. PMID 30652520
- [Background] Wang Y, Coyne K, Sofen H, Santanello N, Currie B, Zhang Z, Nograles K. Qualitative analysis and reproducibility assessment of the Scalp Itch Numeric Rating Scale among patients with moderate to severe plaque psoriasis of the scalp. J Dermatolog Treat. 2019 Dec;30(8):775-783. doi: 10.1080/09546634.2019.1577546. Epub 2019 Mar 5. PMID 30747550
- [Result] Strand V, Fiorentino D, Hu C, Day RM, Stevens RM, Papp KA. Improvements in patient-reported outcomes with apremilast, an oral phosphodiesterase 4 inhibitor, in the treatment of moderate to severe psoriasis: results from a phase IIb randomized, controlled study. Health Qual Life Outcomes. 2013 May 10;11:82. doi: 10.1186/1477-7525-11-82. PMID 23663752
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a 16-week randomized, double-blind, placebo-controlled phase, and a 8-week active treatment phase. At Week 24, subjects may have continued on active treatment by entering a 28-week extension study, total = 52 weeks; At completion of the extension study, subjects may have entered in a long term extension (LTE) for 5 + years.
Pre-assignment Details: Time gaps between the end of one study phase and start of the next phase precluded the continuation of some of the participants in the study.
Groups:
- Placebo: Participants were initially randomized to identically matching placebo (PBO) tablets twice daily (BID) during the Placebo-controlled Phase (Weeks 0-16)
- Apremilast 10mg BID: Participants were initially randomized to apremilast (APR) 10 mg by mouth (PO) BID during the Placebo-controlled Phase (Weeks 0-16).
- Apremilast 20mg BID: Participants were initially randomized to apremilast (APR) 20 mg PO BID during the Placebo-controlled Phase (Weeks 0-16). Also includes those originally randomized to placebo that were re-randomized at Week 16 to APR 20 mg.
- Apremilast 30 mg BID: Participants were initially randomized to apremilast (APR) 30 mg PO BID during the Placebo-controlled Phase (Weeks 0-16). Also includes participants originally randomized to placebo that were re-randomized at Week 16 to APR 30 mg.
- Placebo-Apremilast 20mg BID: Participants who were initially randomized to placebo BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at Week 16 to apremilast 20 mg PO BID and continued dosing with apremilast 20 mg BID during the active treatment phase (Weeks 16-24). At Week 24 (End of core study and beginning of extension study), participants were given the option to enroll into an extension study (PSOR-005E NCT00953875) and continued on the same apremilast dosage they had received at the end of the core study (Weeks 24-52). Participants who elected not to enter into the treatment extension study, completed a 4-week observational follow-up phase of the core study.
- Placebo-Apremilast 30 mg BID: Participants who were initially randomized to placebo BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at Week 16 to apremilast 30 mg PO BID and continued dosing with apremilast 30 mg PO BID during the active treatment phase (Weeks 16-24). At Week 24 (End of core study and beginning of extension study), participants were given the option to enroll into the extension study (PSOR-005E NCT00953875) and continued on the same apremilast dosage they had received at the end of the core study (Weeks 24-52). Participants who elected not to enter into the treatment extension study, completed a 4-week observational follow-up phase of the core study.
Period: Core: Placebo Controlled Phase Week 0-16
Arm/Group | Placebo | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Started | 88 | 89 | 87 | 88 | 0 | 0
Completed | 72 (2 participants completed placebo controlled phase but elected not to continue) | 79 (2 participants completed placebo controlled phase but elected not to continue) | 66 | 70 (3 participants completed placebo controlled phase but elected not to continue) | 0 | 0
Not Completed | 16 | 10 | 21 | 18 | 0 | 0
Not completed — Adverse Event | 5 | 1 | 8 | 10 | 0 | 0
Not completed — Lack of Efficacy | 4 | 3 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 6 | 4 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 3 | 4 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 1 | 1 | 0 | 0
Period: Core: Active Treatment Phase Week 16-24
Arm/Group | Placebo | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Started | 0 (Placebo participants were re-randomized at Week 16 to receive apremilast 20mg or 30mg PO BID.) | 77 (2 participants elected not to continue from previous period) | 66 | 67 (3 participants elected not to continue from previous period) | 34 | 36
Completed | 0 | 65 | 59 | 65 | 33 | 31
Not Completed | 0 | 12 | 7 | 2 | 1 | 5
Not completed — Adverse Event | 0 | 4 | 0 | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 4 | 4 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0
Period: Extension: Active Treatment Week 24-52
Arm/Group | Placebo | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Started | 0 | 47 | 50 | 58 | 27 | 27
Completed Extension and Continued LTE | 0 | 5 | 10 | 10 | 4 | 4
Completed | 0 | 34 (Those dosed APR 10 mg BID in extension study were randomly assigned APR 20 mg or 30 mg BID in LTE) | 33 | 48 | 22 | 19
Not Completed | 0 | 13 | 17 | 10 | 5 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 8 | 10 | 3 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 2 | 2 | 3
Not completed — Lost to Follow-up | 0 | 2 | 5 | 3 | 0 | 1
Not completed — Other | 0 | 0 | 1 | 2 | 0 | 1
Period: LTE Period: Week 52 to 6 Years
Arm/Group | Placebo | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Started | 0 | 0 | 16 (Those dosed APR 10 mg BID in extension study were randomly assigned APR 20 mg or 30 mg BID in LTE) | 17 (Those dosed APR 10 mg BID in extension study were randomly assigned APR 20 mg or 30 mg BID in LTE) | 0 | 0
Completed | 0 | 0 | 4 (Completed = Completed Long Term Extension study) | 5 (Completed = Completed Long Term Extension study) | 0 | 0
Not Completed | 0 | 0 | 12 | 12 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 4 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of all randomized participants.
Groups:
- Placebo: Participants were initially randomized to identically matching placebo (PBO) tablets twice daily BID during the Placebo-controlled Phase (Weeks 0-16).
- Apremilast 10mg BID: Participants were initially randomized to apremilast 10 mg PO BID during the Placebo-controlled Phase (Weeks 0-16).
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Total
Number analyzed (Participants) | 88 | 89 | 87 | 88 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (13.68) | 44.4 (13.96) | 44.6 (12.62) | 44.1 (14.67) | 44.3 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 26 | 32 | 38 | 131
  Male | 53 | 63 | 55 | 50 | 221
Race/Ethnicity, Customized [Number; unit: participants]
  White | 83 | 82 | 82 | 80 | 327
  Black or African American | 1 | 2 | 1 | 2 | 6
  Asian | 4 | 3 | 2 | 4 | 13
  Native Hawaiian/Pacific Islanders | 0 | 0 | 1 | 0 | 1
  American Indian/Alaska Native | 0 | 2 | 0 | 1 | 3
  Other | 0 | 0 | 1 | 1 | 2
Duration of Plaque Psoriasis [Mean (Standard Deviation); unit: years] — A diagnosis of chronic plaque psoriasis for ≥ 6 months was required prior to screening. Those with moderate to severe plaque psoriasis must have had a Psoriasis Area Severity Index (PASI) score ≥ 12, (PASI was a measure of psoriatic disease severity taking into account lesion characteristics (erythema, thickness, and scaling) and degree of skin and body surface area involvement (BSA) on defined anatomical regions), BSA ≥ 10. Duration of plaque psoriasis was calculated from the date of diagnosis to the date of informed consent. The dates of diagnosis were not available for some participants
  years | 19.61 (11.632) | 18.01 (12.366) | 19.51 (12.151) | 19.18 (12.015) | 18.99 (12.004)

OUTCOME MEASURES:

1. Primary Outcome: Core Study: Percentage of Participants Who Achieved a 75% Improvement (Response) in Psoriasis Area and Severity Index (PASI) at Week 16
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 and Week 16
Population: The intent-to-treat (ITT) population = all randomized participants. Last observation carried forward (LOCF) method was used for imputing missing values
Measure: Number; unit: percentage of participants
Groups:
- Placebo BID: Participants were initially randomized to placebo PO BID during the Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 88 | 89 | 87 | 88
percentage of participants | 5.7 | 11.2 | 28.7 | 40.9
Statistical Analysis 1: Comparison: Placebo BID vs Apremilast 10mg BID; Test type: Superiority or Other; p = 0.1846, Chi-squared; Risk Difference (RD) = 5.6, 95% CI 2-sided [-2.6 to 13.7]
Statistical Analysis 2: Comparison: Placebo BID vs Apremilast 20mg BID; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 23.1, 95% CI 2-sided [12.4 to 33.7]
Statistical Analysis 3: Comparison: Placebo BID vs Apremilast 30 mg BID; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 35.2, 95% CI 2-sided [23.9 to 46.6]

2. Secondary Outcome: Core Study: Percentage of Participants Who Achieved a 75% Improvement (Response) in PASI Score at Week 24
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 24. The improvement in PASI score was used as a measure of efficacy.The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head,trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 24
Population: Intent to Treat; Placebo participants re-randomized at Week 16; End of Period = Last observation carried forward in the period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apremilast 10mg BID: Participants who were initially randomized to apremilast 10mg PO BID during the Placebo-controlled Phase (Weeks 0-16) remained on APR 10 mg BID PO during the Active Treatment Phase (Weeks 16-24).
- PBO-Apremilast 20mg BID: Participants who were initially randomized to placebo BID PO during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at week 16 to apremilast 20 mg PO BID and continued dosing with apremilast 20 mg PO BID during the active treatment phase (Weeks 16-24).
- PBO-Apremilast 30 mg BID: Participants who were initially randomized to placebo BID PO during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at Week 16 to apremilast 30 mg PO BID and continued dosing with apremilast 30 mg BID during the active treatment phase (Weeks 16-24).
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | PBO-Apremilast 20mg BID | PBO-Apremilast 30 mg BID
Number analyzed (Participants) | 89 | 87 | 88 | 34 | 36
percentage of participants | 18.0 [10.6 to 27.5] | 26.4 [17.6 to 37.0] | 39.8 [29.5 to 50.8] | 41.2 [24.6 to 59.3] | 44.4 [27.9 to 61.9]

3. Secondary Outcome: Core Study: Percentage of Participants Who Achieved a 50% Improvement (Response) in PASI Score at Week 16
Description: PASI-50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy The PASI score was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 88 | 89 | 87 | 88
percentage of participants | 25.0 | 38.2 | 47.1 | 60.2
Statistical Analysis 1: Comparison: Placebo BID vs Apremilast 10mg BID; Test type: Superiority or Other; p = 0.0590, Chi-squared; Risk Difference (RD) = 13.2, 95% CI 2-sided [-0.4 to 26.8]
Statistical Analysis 2: Comparison: Placebo BID vs Apremilast 20mg BID; Test type: Superiority or Other; p = 0.0023, Chi-squared; Risk Difference (RD) = 22.1, 95% CI 2-sided [8.3 to 36.0]
Statistical Analysis 3: Comparison: Placebo BID vs Apremilast 30 mg BID; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 35.2, 95% CI 2-sided [21.6 to 48.9]

4. Secondary Outcome: Core Study: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score at Week 24
Description: PASI-50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score at Week 24. The improvement in PASI score was used as a measure of efficacy. The PASI score was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apremilast 10mg BID: Participants who were initially randomized to apremilast 10 mg PO BID during the Placebo-controlled Phase (Weeks 0-16) remained on apremilast 10 mg BID during the Active Treatment Phase (Weeks 16-24).
- Apremilast 20mg: Participants who were initially randomized to apremilast 20 mg PO BID during the Placebo-controlled Phase (Weeks 0-16) remained on apremilast 20 mg BID during the Active Treatment Phase (Weeks 16-24).
- PBO-Apremilast 30 mg BID: Participants who were initially randomized to placebo BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at week 16 to apremilast 30 mg PO BID and continued dosing with apremilast 30 mg BID during the active treatment phase (Weeks 16-24).
Arm/Group | Apremilast 10mg BID | Apremilast 20mg | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | PBO-Apremilast 30 mg BID
Number analyzed (Participants) | 89 | 87 | 88 | 34 | 36
percentage of participants | 38.2 [28.1 to 49.1] | 49.4 [38.5 to 60.4] | 65.9 [55.0 to 75.7] | 61.8 [43.6 to 77.8] | 75.0 [57.8 to 87.9]

5. Secondary Outcome: Core Study: Percentage of Participants Who Achieved a 90% Improvement (Response) From Baseline in the PASI Score at Week 16
Description: PASI-90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. The PASI score was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 88 | 89 | 87 | 88
percentage of participants | 1.1 | 4.5 | 9.2 | 11.4
Statistical Analysis 1: Comparison: Placebo BID vs Apremilast 10mg BID; Test type: Superiority or Other; p = 0.1776, Chi-squared; Risk Difference (RD) = 3.4, 95% CI 2-sided [-1.5 to 8.2]
Statistical Analysis 2: Comparison: Placebo BID vs Apremilast 20mg BID; Test type: Superiority or Other; p = 0.0158, Chi-squared; Risk Difference (RD) = 8.1, 95% CI 2-sided [1.6 to 14.5]
Statistical Analysis 3: Comparison: Placebo BID vs Apremilast 30 mg BID; Test type: Superiority or Other; p = 0.0051, Chi-squared; Risk Difference (RD) = 10.2, 95% CI 2-sided [3.2 to 17.2]

6. Secondary Outcome: Core Study: Percentage of Participants Who Achieved a 90% Improvement (Response) in the PASI Score at Week 24
Description: PASI-90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 24. The improvement in PASI score was used as a measure of efficacy..The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling were scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions was scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apremilast 10mg: Participants who were initially randomized to apremilast 10 mg PO BID during the Placebo-controlled Phase (Weeks 0-16) remained on apremilast 10 mg BID during the Active Treatment Phase (Weeks 16-24).
- Apremilast 30 mg: Participants who were initially randomized to apremilast 30 mg PO BID during the Placebo-controlled Phase (Weeks 0-16) remained on apremilast 30 mg BID during the Active Treatment Phase (Weeks 16-24).
- PBO-Apremilast 20mg BID: Participants who were initially randomized to placebo BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at week 16 to apremilast 20 mg BID and continued dosing with apremilast 20 mg BID during the active treatment phase (Weeks 16-24).
Arm/Group | Apremilast 10mg | Apremilast 20mg | Apremilast 30 mg | PBO-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 89 | 87 | 88 | 34 | 36
percentage of participants | 4.5 [1.2 to 11.1] | 8.0 [3.3 to 15.9] | 14.8 [8.1 to 23.9] | 14.7 [5.0 to 31.1] | 16.7 [6.4 to 32.8]

7. Secondary Outcome: Core Study: Percentage of Participants Who Achieved a 100% Improvement (Response) in the PASI Score at Week 16
Description: A participant was classified as having achieved a PASI-100 response if the PASI score was reduced by at least 100% from baseline. The PASI score was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 16
Population: The PASI 100 was not defined and analyzed since there were too few such participants.
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Core Study: Percentage of Participants Who Achieved a 100% Improvement (Response) in the PASI Score at Week 24
Description: as for outcome 7
Time Frame: Week 0 to Week 24
Population: The PASI 100 was not defined and analyzed since there were too few such participants.
Groups:
- Apremilast 10mg BID: Participants who were initially randomized to APR 10 mg PO BID during the Placebo-controlled Phase (Weeks 0-16) remained on apremilast 10 mg BID during the Active Treatment Phase (Weeks 16-24).
- PBO-Apremilast 20mg BID: Participants who were initially randomized to identically matching placebo BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at week 16 to apremilast 20 mg tablets BID and continued dosing with apremilast 20 mg BID during the active treatment phase (Weeks 16-24).
- PBO-Apremilast 30 mg BID: Participants who were initially randomized to identically matching placebo BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at week 16 to apremilast 30 mg PO BID and continued dosing with apremilast 30 mg BID during the active treatment phase (Weeks 16-24).
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | PBO-Apremilast 20mg BID | PBO-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Core Study: Time to Achieve a PASI-100 Response During the Placebo Controlled Phase
Description: For PASI-100 responders in the placebo-controlled period weeks 0-16, time to achieve PASI-100 was the time interval, inclusive, between the date of randomization (day 1) and the date of the first assessment where PASI-90 was achieved.
Time Frame: Weeks 0 to 16
Population: Time to achieve PASI 100 was not defined or analyzed as there were too few participants.
Groups:
- Placebo BID: Participants were initially randomized to identically matching placebo (PBO) tablets twice daily (BID) during the Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Core Study: Percent Change From Baseline in PASI Score at Week 16
Description: The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling were scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions was scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) was multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. The values for each anatomic region were summed to yield the PASI score.
Time Frame: Week 0 to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Placebo BID: Participants were initially randomized to placebo PO BID during the Placebo-controlled Phase (Weeks 0-16). .
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 88 | 87 | 82 | 87
Percent change | -20.3 (3.98) | -34.0 (4.00) | -45.4 (4.12) | -53.2 (4.00)
Statistical Analysis 1: Comparison: Placebo BID vs Apremilast 10mg BID; Test type: Superiority or Other; p = 0.0156, ANCOVA; Analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Least Square Mean Difference = -13.7, 95% CI 2-sided [-24.8 to -2.6]
Statistical Analysis 2: Comparison: Placebo BID vs Apremilast 20mg BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of covariance model with treatment group as a factor and the baseline value as a covariate; LS Mean Difference = -25.1, 95% CI 2-sided [-36.4 to -13.9]
Statistical Analysis 3: Comparison: Placebo BID vs Apremilast 30 mg BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of covariance model with treatment group as a factor and the baseline value as a covariate; LS Mean Difference = -32.9, 95% CI 2-sided [-44.0 to -21.7]

11. Secondary Outcome: Core Study: Percent Change From Baseline in PASI Score at Week 24
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling were scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions was scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) was multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. The values for each anatomic region were summed to yield the PASI score
Time Frame: Week 0 to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- PBO-Apremilast 20mg BID: Participants who were initially randomized to placebo BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at week 16 to apremilast 20 mg PO BID and continued dosing with apremilast 20 mg BID during the active treatment phase (Weeks 16-24
- PBO-Apremilast 30 mg BID: Participants who were initially randomized to placebo BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at week 16 to apremilast 30 mg PO BID and continued dosing with apremilast 30 mg BID during the active treatment phase (Weeks 16-24.
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | PBO-Apremilast 20mg BID | PBO-Apremilast 30 mg BID
Number analyzed (Participants) | 87 | 82 | 87 | 34 | 36
percent change | -36.3 (36.03) | -46.5 (36.08) | -56.8 (34.99) | -61.7 (25.35) | -61.7 (32.67)

12. Other Pre Specified Outcome: Core Study: Percentage of Participants With a Static Physician Global Assessment (sPGA) Greater Than 2 at Baseline Who Achieved a Score of 0 or 1 at Week 16
Description: The sPGA was a measure of psoriasis disease severity at the time of evaluation by the investigator. It does not compare assessments across visits or rely on investigator recall of prior disease severity. The sPGA was a 6-point scale ranging from 0 (clear, except for residual discoloration) to 5 (severe; majority of plaques have severe thickness, erythema, and scaling). The investigator examined all of the lesions on the participant and assigned a score ranging from 0 to 5 for thickness, erythema and degree of scaling . Scores for thickness, erythema and scaling are then summed and the mean of these 3 scores equaled the overall sPGA score. Fractional values for the sPGA were rounded to the next highest integer (eg, a score of 3.5 was rounded to 4, 3.4 was rounded to 3). A lower sPGA score was associated with less severe disease
Time Frame: Week 0 to Week 16
Population: Intent to Treat; Last observation carried forward (LOCF) method was used for imputing missing values
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants were initially randomized to placebo PO BID during the Placebo-controlled Phase (Weeks 0-16)
- Apremilast 10mg: Participants were initially randomized to apremilast 10 mg PO BID during the Placebo-controlled Phase (Weeks 0-16).
- Apremilast 20mg: Participants were initially randomized to apremilast 20 mg PO BID during the Placebo-controlled Phase (Weeks 0-16).
- Apremilast 30 mg: Participants were initially randomized to apremilast 30 mg PO BID during the Placebo-controlled Phase (Weeks 0-16).
Arm/Group | Placebo | Apremilast 10mg | Apremilast 20mg | Apremilast 30 mg
Number analyzed (Participants) | 87 | 86 | 80 | 83
percentage of participants | 12.6 | 10.5 | 25.0 | 33.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 10mg; Test type: Superiority or Other; p = 0.6541, Chi-squared; Risk Difference (RD) = -2.2, 95% CI 2-sided [-11.7 to 7.3]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20mg; Test type: Superiority or Other; p = 0.0402, Chi-squared; Risk Difference (RD) = 12.4, 95% CI 2-sided [0.6 to 24.1]
Statistical Analysis 3: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0011, Chi-squared; Risk Difference (RD) = 21.1, 95% CI 2-sided [8.8 to 33.4]

13. Other Pre Specified Outcome: Core Study: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of 0 or 1 at Week 24
Description: as for outcome 12
Time Frame: Week 0 and Week 24
Population: Intent to Treat; Placebo participants re-randomized at Week 16; Last observation carried forward in the period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo-Apremilast 20 mg BID: Participants who were initially randomized to placebo PO BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at week 16 to apremilast 20 mg PO BID and continued dosing with apremilast 20 mg BID during the active treatment phase (Weeks 16-24).
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20 mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 89 | 87 | 88 | 34 | 36
percentage of participants | 13.5 [7.2 to 22.4] | 24.1 [15.6 to 34.5] | 34.1 [24.3 to 45.0] | 41.2 [24.6 to 59.3] | 50.0 [32.9 to 67.1]

14. Secondary Outcome: Core Study: Shift Change (1 or More Points on a 0 to 5 Point Scale) in Static Physician Global Assessment (sPGA) at Week 16
Description: Physician Global Assessment (sPGA) was a measure of psoriasis disease severity at the time of evaluation by the investigator. It does not compare assessments across visits or rely on investigator recall of prior disease severity. The sPGA is a 6-point scale ranging from 0 (clear, except for residual discoloration) to 5 (severe; majority of plaques have severe thickness, erythema, and scaling). The investigator examined all of the lesions on the participant and assigned a score ranging from 0 to 5 for thickness, erythema and degree of scaling. Scores for thickness, erythema and scaling are then summed and the mean of these 3 scores equaled the overall sPGA score. Fractional values for the sPGA were rounded to the next highest integer (eg, a score of 3.5 was rounded to 4, 3.4 was rounded to 3).
Time Frame: Week 0 to Week 16
Population: The Shift change in sPGA was not defined and analyzed. A response defined as achieving sPGA score 0 or 1 with at least 2 points reduction from baseline was a more meaningful clinical endpoint. See other pre-specified outcome measures.
Groups:
- Apremilast 10mg BID: Participants were initially randomized to apremilast (APR) 10 mg tablets BID during the Placebo-controlled Phase (Weeks 0-16).
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Core Study: Shift Change (1 or More Points on a 0 to 5 Point Scale) in Static Physician Global Assessment (sPGA) at Week 24
Description: as for outcome 14
Time Frame: Week 0 to Week 24
Population: The Shift change in sPGA was not defined and analyzed. A response defined as achieving sPGA score 0 or 1 with at least 2 points reduction from baseline was a more meaningful clinical endpoint.
Groups:
- Placebo-Apremilast 20 mg BID: Participants who were initially randomized to placebo BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at week 16 to apremilast 20 mg PO BID and continued dosing with apremilast 20 mg BID during the active treatment phase (Weeks 16-24).
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20 mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Core Study: Percent Change From Baseline in the Percent of Affected Body Surface Area (BSA) During the Placebo Controlled Phase
Description: The overall BSA affected by psoriasis was estimated by comparison of the size of the affected area to the palm area of the participant's hand (entire palmar surface or "handprint"), which equates to approximately 1% of total BSA.
Time Frame: Week 0 to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 88 | 87 | 82 | 87
percent change | -8.0 (4.58) | -28.3 (4.60) | -38.0 (4.74) | -50.4 (4.63)
Statistical Analysis 1: Comparison: Placebo BID vs Apremilast 10mg BID; Test type: Superiority or Other; p = 0.0020, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; LS Mean Difference = -20.2, 95% CI 2-sided [-33.0 to -7.5]
Statistical Analysis 2: Comparison: Placebo BID vs Apremilast 20mg BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; LS Mean Difference = -29.9, 95% CI 2-sided [-42.9 to -17.0]
Statistical Analysis 3: Comparison: Placebo BID vs Apremilast 30 mg BID; Test type: Superiority or Other; p < 0.0001, ANCOVA — Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; LS Mean Difference = -42.4, 95% CI 2-sided [-55.2 to -29.5]

17. Secondary Outcome: Core Study: Percent Change From Baseline in the Percent of Affected Body Surface Area (BSA) During the Active Treatment Phase at Week 24
Description: as for outcome 16
Time Frame: Week 0 to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20 mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 87 | 82 | 87 | 34 | 36
percent change | -28.1 (46.78) | -40.6 (43.71) | -54.0 (37.32) | -52.5 (37.35) | -54.2 (42.08)

18. Secondary Outcome: Core Study: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI was a validated, self-administered, 10-item questionnaire that measures the impact of skin disease on subjects' quality of life, based on recall over the past week. Domains include symptoms, feelings, daily activities, social, leisure, work or studying, personal relationships and treatment. Each question on the extent of the impact of skin disease was answered on a scale of 0 (not at all) to 3 (very much); the total DLQI score ranged from 0 to 30. A DLQI score greater than 10 is indicative of severe psoriasis.
Time Frame: Week 0 to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 83 | 87 | 78 | 83
units on a scale | -1.9 (0.63) | -3.2 (0.62) | -5.9 (0.65) | -4.4 (0.63)
Statistical Analysis 1: Comparison: Placebo BID vs Apremilast 10mg BID; Test type: Superiority or Other; p = 0.1322, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Difference in LS Means = -1.3, 95% CI 2-sided [-3.1 to 0.4]
Statistical Analysis 2: Comparison: Placebo BID vs Apremilast 20mg BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Difference in LS Means = -4.1, 95% CI 2-sided [-5.9 to -2.3]
Statistical Analysis 3: Comparison: Placebo BID vs Apremilast 30 mg BID; Test type: Superiority or Other; p = 0.0047, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Difference in LS Means = -2.6, 95% CI 2-sided [-4.3 to -0.8]

19. Secondary Outcome: Core Study: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 24
Description: as for outcome 18
Time Frame: Week 0 to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo-Apremilast (APR) 20 mg BID: Participants who were initially randomized to placebo PO BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at Week 16 to apremilast 20 mg PO BID and continued dosing with apremilast 20 mg BID during the active treatment phase (Weeks 16-24).
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast (APR) 20 mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 87 | 78 | 83 | 34 | 36
units on a scale | -3.4 (6.40) | -6.2 (6.53) | -4.9 (5.18) | -6.4 (6.64) | -5.4 (5.32)

20. Secondary Outcome: Core Study: Change From Baseline in the Medical Outcome Study Short Form 36-Item Health Survey (SF-36), Version 2; Mental Component Summary Score at Week 16
Description: The SF-36 was a 36-item general health status instrument and consists of 8 scales: physical function (PF), role limitations-physical (RP), vitality (VT), general health perceptions (GH), bodily pain (BP), social function (SF), role limitations-emotional (RE), and mental health (MH). Scale scores range from 0 to 100, with higher scores indicating better health. Two overall summary scores were obtained - a Physical Component Summary score (PCS) and a Mental Component Summary score (MCS). Scores from the 8 scales, PCS and MCS were transformed to the norm-based scores using weights from U.S. general population, with 50 as the average and 10 as the standard deviation, higher scores indicating better health. For norm based scores, change from baseline were calculated for the 8 scales and the two summary scales, where change = visit value - baseline value.
Time Frame: Week 0 to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 83 | 87 | 78 | 84
units on a scale | -0.6 (0.89) | 2.8 (0.87) | 2.9 (0.92) | 3.0 (0.89)
Statistical Analysis 1: Comparison: Placebo BID vs Apremilast 10mg BID; Test type: Superiority or Other; p = 0.0078, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Difference in LS Means = 3.3, 95% CI 2-sided [0.9 to 5.8]
Statistical Analysis 2: Comparison: Placebo BID vs Apremilast 20mg BID; Test type: Superiority or Other; p = 0.0068, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Difference in LS Means = 3.5, 95% CI 2-sided [1.0 to 6.0]
Statistical Analysis 3: Comparison: Placebo BID vs Apremilast 30 mg BID; Test type: Superiority or Other; p = 0.0045, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Difference in LS Means = 3.6, 95% CI 2-sided [1.1 to 6.1]

21. Secondary Outcome: Core Study: Change From Baseline in the Medical Outcome Study Short Form 36-Item Health Survey (SF-36), Version 2; Physical Component Summary Score at Week 16
Description: as for outcome 20
Time Frame: Week 0 to week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 83 | 87 | 78 | 84
units on a scale | 0.7 (0.80) | 1.3 (0.78) | 2.1 (0.83) | 0.8 (0.80)
Statistical Analysis 1: Comparison: Placebo BID vs Apremilast 10mg BID; Test type: Superiority or Other; p = 0.6097, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Difference in LS Means = 0.6, 95% CI 2-sided [-1.6 to 2.8]
Statistical Analysis 2: Comparison: Placebo BID vs Apremilast 20mg BID; Test type: Superiority or Other; p = 0.2424, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Difference in LS Means = 1.3, 95% CI 2-sided [-0.9 to 3.6]
Statistical Analysis 3: Comparison: Placebo BID vs Apremilast 30 mg BID; Test type: Superiority or Other; p = 0.9528, ANCOVA; Based on an analysis of covariance model with treatment group as a factor and the baseline value as a covariate; Difference in LS Means = 0.1, 95% CI 2-sided [-2.2 to 2.3]

22. Secondary Outcome: Core Study: Change From Baseline in the Medical Outcome Study Short Form 36-Item Health Survey (SF-36), Version 2; Mental Component Summary Score at Week 24
Description: as for outcome 20
Time Frame: Week 0 to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PBO-Apremilast 20mg BID: Participants who were initially randomized to placebo PO BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at Week 16 to apremilast 20 mg PO BID and continued dosing with apremilast 20 mg BID during the active treatment phase (Weeks 16-24).
- PBO-Apremilast 30 mg BID: Participants who were initially randomized to placebo PO BID during the Placebo-controlled Phase (Weeks 0-16) were re-randomized at Week 16 to apremilast 30 mg PO BID and continued dosing with apremilast 30 mg BID during the active treatment phase (Weeks 16-24).
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | PBO-Apremilast 20mg BID | PBO-Apremilast 30 mg BID
Number analyzed (Participants) | 87 | 78 | 84 | 34 | 36
units on a scale | 2.8 (9.16) | 3.9 (9.56) | 2.9 (10.22) | 2.8 (10.96) | 0.5 (9.17)

23. Secondary Outcome: Core Study: Change From Baseline in the Medical Outcome Study Short Form 36-Item Health Survey (SF-36), Version 2 Physical Component Summary Score at Week 24
Description: as for outcome 20
Time Frame: Week 0 to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | PBO-Apremilast 20mg BID | PBO-Apremilast 30 mg BID
Number analyzed (Participants) | 87 | 78 | 84 | 34 | 36
units on a scale | 1.1 (6.42) | 2.3 (8.29) | 1.0 (7.72) | 2.5 (9.34) | 2.7 (8.24)

24. Secondary Outcome: Core Study: Area Under the Plasma Concentration-time Curve (AUC0-8)
Description: Area under the concentration versus time curve from time 0 (pre-dose) to 8 hours, calculated using the linear trapezoid rule.
Time Frame: Week 14; Predose, 0.5, 1, 2, 3, 4, and 8 hours after the morning dose of apremilast
Population: Pharmacokinetic population; samples were not obtained from participants who were randomized to placebo
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Apremilast 10mg BID: Participants were initially randomized to placebo PO BID during the Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 7 | 5 | 3
ng*h/mL | 1008 (35.8) | 1591 (56.9) | 3467 (20.8)

25. Secondary Outcome: Core Study: Area Under the Plasma Concentration-time Curve (AUC0-8)
Description: Area under the concentration versus time curve from time 0 (pre-dose) to 8 hours, calculate using the linear trapezoid rule.
Time Frame: Week 24
Population: Pharmacokinetic population; samples were not obtained from participants who were randomized to placebo.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Apremilast 10mg | Apremilast 20mg | Apremilast 30 mg
Number analyzed (Participants) | 5 | 4 | 3
ng*h/mL | 1200 (44.6) | 1257 (47.1) | 3477 (29.3)

26. Secondary Outcome: Core Study: Peak; (Maximum) Plasma Concentration (Cmax) of Apremilast
Description: The maximum observed plasma concentration of apremilast observed at Week 14 (steady-state Cmax)
Time Frame: Week 14; Predose, 0.5, 1, 2, 3, 4, and 8 hours after the morning dose of apremilast
Population: Pharmacokinetic population; samples were not obtained from participants who were randomized to placebo
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 7 | 5 | 3
ng/mL | 209 (27.9) | 298 (48.3) | 637 (18.7)

27. Secondary Outcome: Core Study: Peak; (Maximum) Plasma Concentration (Cmax) of Apremilast
Description: The maximum observed plasma concentration of apremilast observed at Week 24 (steady-state Cmax)
Time Frame: Week 24
Population: Pharmacokinetic population; samples were not obtained from participants who were randomized to placebo.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 3
ng/mL | 238 (45.2) | 236 (39.7) | 670 (20.4)

28. Secondary Outcome: Core Study: Time to Maximum Plasma Concentration of Drug (Tmax)
Description: Time to achieve maximum plasma concentration (Cmax) observed at Week 14 (Time to achieve steady-state Tmax)
Time Frame: Week 14; Predose, 0.5, 1, 2, 3, 4, and 8 hours after the morning dose of apremilast
Population: Pharmacokinetic population; samples were not obtained from participants who were randomized to placebo
Measure: Median (Full Range); unit: hours
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 7 | 5 | 3
hours | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 1.00 [1.00 to 2.00]

29. Secondary Outcome: Core Study: Time to Maximum Plasma Concentration of Drug (Tmax)
Description: Time to achieve maximum plasma concentration (tmax) observed at Week 24 (Time to achieve steady-state Tmax)
Time Frame: Week 24
Population: Pharmacokinetic population; samples were not obtained from participants who were randomized to placebo
Measure: Median (Full Range); unit: hours
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 3
hours | 1.00 [1.00 to 3.00] | 1.50 [1.00 to 4.00] | 1.00 [0.500 to 1.00]

30. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 75% Improvement (Response) in the PASI Score at Week 52
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 52. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 52
Population: Includes participants who entered the extension study; LOCF was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apremilast 10mg BID: Participants who were initially randomized to apremilast 10 mg PO BID during the Placebo-controlled Phase (Weeks 0-16) remained on apremilast 10 mg BID during the Active Treatment Phase (Weeks 16-24) and during the extension study (Weeks 24-52).
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 14.9 [6.2 to 28.3] | 22.0 [11.5 to 36.0] | 36.2 [24.0 to 49.0] | 37.0 [19.4 to 57.6] | 33.3 [16.5 to 54.0]

31. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 75% Improvement (Response) in the PASI Score at Week 32
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 32 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 32
Population: Includes participants who entered the extension study; Intent to Treat; Non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 27.7 [15.6 to 42.6] | 38.0 [24.7 to 52.8] | 46.6 [33.3 to 60.1] | 33.3 [16.5 to 54.0] | 55.6 [35.3 to 74.5]

32. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 75% Improvement (Response) in the PASI Score at Week 40
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 40 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 40
Population: Includes participants who entered the extension study; Intent to Treat; Non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 21.3 [10.7 to 35.7] | 28.0 [16.2 to 42.5] | 34.5 [22.5 to 48.1] | 37.0 [19.4 to 57.6] | 44.4 [25.5 to 64.7]

33. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score at Week 32
Description: PASI-50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score at Week 32 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 32
Population: Includes participants who entered the extension study; Intent to Treat; Non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 57.4 [42.2 to 71.7] | 72.0 [57.5 to 83.8] | 86.2 [74.6 to 93.9] | 74.1 [53.7 to 88.9] | 74.1 [53.7 to 88.9]

34. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score at Week 40
Description: PASI-50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score at Week 16 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 40
Population: Includes participants who entered the extension study; Intent to Treat; Non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 48.9 [34.1 to 63.9] | 62.0 [47.2 to 75.3] | 82.8 [70.6 to 91.4] | 63.0 [42.4 to 80.6] | 66.7 [46.0 to 83.5]

35. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score at Week 52
Description: PASI-50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score at Week 52 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 52
Population: Includes participants who entered the extension study; Intent to Treat; Non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 42.6 [28.3 to 57.8] | 48.0 [33.7 to 62.6] | 72.4 [59.1 to 83.6] | 55.6 [35.3 to 74.5] | 48.1 [28.7 to 68.1]

36. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 90% Improvement (Response) in the PASI Score at Week 32
Description: PASI-90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 32 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 32
Population: Includes participants who entered the extension study; Intent to Treat; Non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 10.6 [3.5 to 23.1] | 14.0 [5.8 to 26.7] | 19.0 [9.9 to 31.4] | 18.5 [6.3 to 38.1] | 25.9 [11.1 to 46.3]

37. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 90% Improvement (Response) in the PASI Score at Week 40
Description: PASI-90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 40 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 40
Population: Includes participants who entered the extension study; Intent to Treat; Non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 8.5 [2.4 to 20.4] | 14.0 [5.8 to 26.7] | 17.2 [8.6 to 29.4] | 18.5 [6.3 to 38.1] | 22.2 [8.6 to 42.3]

38. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 90% Improvement (Response) in the PASI Score at Week 52
Description: PASI-90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 52 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Week 52
Population: Includes participants who entered the extension study; Intent to Treat; Non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 4.3 [0.5 to 14.5] | 10.0 [3.3 to 21.8] | 13.8 [6.1 to 25.4] | 14.8 [4.2 to 33.7] | 11.1 [2.4 to 29.2]

39. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 100% Improvement (Response) in the PASI Score at Week 32
Description: as for outcome 7
Time Frame: Week 0 to Week 32
Population: The PASI 100 was not defined and analyzed since there were too few such participants.
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 100% Improvement (Response) in the PASI Score at Week 40
Description: as for outcome 7
Time Frame: Week 0 to Week 40
Population: The PASI 100 was not defined and analyzed since there were too few such participants.
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Extension Study: Percentage of Participants Who Achieved a 100% Improvement (Response) in the PASI Score at Week 52
Description: as for outcome 7
Time Frame: Week 0 to Week 52
Population: The PASI 100 was not defined and analyzed since there were too few such participants.
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Extension Study: Time to Achieve PASI-75 During the Extension Study
Description: For PASI-75 responders in the extension study, time to achieve PASI-75 was defined as the time interval, inclusive between the date of randomization (Day 1) and the date of the first assessment where PASI-75 was achieved.
Time Frame: Week 0 to Week 52
Population: Time to achieve PASI-75 score was not defined and analyzed as there were too few such participants who did not achieve responses in the core study but achieved in the extension study
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

43. Secondary Outcome: Extension Study: Time to Achieve PASI-50 During the Extension Study
Description: For PASI-50 responders in the extension study, time to achieve PASI-50 was defined as the time interval, inclusive between the date of randomization (Day 1) and the date of the first assessment where PASI-50 was achieved.
Time Frame: Week 0 to Week 52
Population: Time to achieve PASI-50 score was not defined and analyzed as there were too few such participants who did not achieve responses in the core study but achieved in the extension study
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Extension Study: Time to Achieve PASI-90 During the Extension Study
Description: For PASI-90 responders in the extension study, time to achieve PASI-90 was defined as the time interval, inclusive between the date of randomization (Day 1) and the date of the first assessment where PASI-90 was achieved.
Time Frame: Week 0 to Extension study
Population: Time to achieve PASI-90 score was not defined and analyzed as there were too few such participants who did not achieve responses in the core study but achieved in the extension study
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

45. Secondary Outcome: Extension Study: Time to Achieve PASI-100 During the Extension Study
Description: For PASI-100 responders in the extension study, time to achieve PASI-100 was defined as the time interval, inclusive between the date of randomization (Day 1) and the date of the first assessment where PASI-100 was achieved.
Time Frame: Week 0 to Extension Study
Population: Time to achieve PASI-100 score was not defined and analyzed as there were too few such participants who did not achieve responses in the core study but achieved in the extension study
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

46. Other Pre Specified Outcome: Extension Study: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of 0 or 1 at Week 32
Description: as for outcome 12
Time Frame: Week 0 to Week 32
Population: Includes participants who entered the extension study; Intent to Treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 23.4 [12.3 to 38.0] | 26 [14.6 to 40.3] | 44.8 [31.7 to 58.5] | 33.3 [16.5 to 54.0] | 59.3 [38.8 to 77.6]

47. Other Pre Specified Outcome: Extension Study: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of 0 or 1 at Week 40
Description: The sPGA was a measure of psoriasis disease severity at the time of evaluation by the investigator. It does not compare assessments across visits or rely on investigator recall of prior disease severity. The sPGA was a 6-point scale ranging from 0 (clear, except for residual discoloration) to 5 (severe; majority of plaques have severe thickness, erythema, and scaling). The investigator examined all of the lesions on the participant and assigned a score ranging from 0 to 5 for thickness, erythema and degree of scaling . Scores for thickness, erythema and scaling are then summed and the mean of these 3 scores equaled the overall sPGA score. Fractional values for the sPGA were rounded to the next highest integer (eg, a score of 3.5 was rounded to 4, 3.4 was rounded to 3). A lower sPGA score was associated with less disease.
Time Frame: Week 0 to Week 40
Population: Includes participants who entered the extension study; Intent to Treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 23.4 [12.3 to 38.0] | 18.0 [8.6 to 31.4] | 29.3 [18.1 to 42.7] | 29.6 [13.8 to 50.2] | 37.0 [19.4 to 57.6]

48. Other Pre Specified Outcome: Extension Study: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of 0 or 1 at Week 52
Description: as for outcome 12
Time Frame: Week 0 to Week 52
Population: Includes participants who entered the extension study; LOCF was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 47 | 50 | 58 | 27 | 27
percentage of participants | 12.8 [4.8 to 25.7] | 10.0 [3.3 to 21.8] | 22.4 [12.5 to 35.3] | 33.3 [16.5 to 54.0] | 22.2 [8.6 to 42.3]

49. Secondary Outcome: Extension Study: Percent Change in PASI Score at Week 32
Description: as for outcome 11
Time Frame: Week 0 to Week 32
Population: Includes participants who entered the extension study and had PASI assessment at Week 32; Intent to Treat
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 43 | 48 | 55 | 26 | 26
percent change | -51.0 (34.10) | -63.1 (27.01) | -72.7 (20.97) | -64.0 (25.16) | -69.2 (27.60)

50. Secondary Outcome: Extension Study: Percent Change in PASI Score at Week 40
Description: as for outcome 11
Time Frame: Week 0 to Week 40
Population: Includes participants who entered the extension study and had PASI assessment at Week 40; Intent to Treat;
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 36 | 40 | 51 | 24 | 21
percent change | -55.9 (29.63) | -63.3 (27.26) | -71.1 (18.91) | -64.5 (27.05) | -71.7 (24.53)

51. Secondary Outcome: Extension Study: Percent Change in PASI Score at Week 52
Description: as for outcome 11
Time Frame: Week 0 to Week 52
Population: Includes participants who entered the extension study and had PASI assessment at Week 52; Intent to Treat;
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 34 | 34 | 49 | 22 | 19
percent change | -55.1 (23.50) | -58.9 (30.65) | -65.3 (29.86) | -62.7 (29.49) | -62.0 (28.28)

52. Secondary Outcome: Extension Study: Shift Change (1 or More Points on a 0 to 5 Point Scale) in Static Physician Global Assessment (sPGA) at Week 32
Description: Physician Global Assessment (sPGA) was a measure of psoriasis disease severity at the time of evaluation by the investigator. It does not compare assessments across visits or rely on investigator recall of prior disease severity. The sPGA is a 6-point scale ranging from 0 (clear, except for residual discoloration) to 5 (severe; majority of plaques have severe thickness, erythema, and scaling). The investigator examined all of the lesions on the subject and assigned a score ranging from 0 to 5 for thickness, erythema and degree of scaling. Scores for thickness, erythema and scaling are then summed and the mean of these 3 scores equaled the overall sPGA score. Fractional values for the sPGA were rounded to the next highest integer (eg, a score of 3.5 was rounded to 4, 3.4 was rounded to 3).
Time Frame: Week 0 to Week 32
Population: The Shift change in sPGA was not defined and analyzed. A response defined as achieving sPGA score 0 or 1 with at least 2 points reduction from baseline was a more meaningful clinical endpoint. See pre-specified outcome measures.
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

53. Secondary Outcome: Extension Study: Shift Change (1 or More Points on a 0 to 5 Point Scale) in Static Physician Global Assessment (sPGA) at Week 40
Description: as for outcome 52
Time Frame: Week 0 to Week 40
Population: as for outcome 52
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

54. Secondary Outcome: Extension Study: Shift Change (1 or More Points on a 0 to 5 Point Scale) in Static Physician Global Assessment (sPGA) at Week 52
Description: as for outcome 52
Time Frame: Week 0 to Week 52
Population: as for outcome 52
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

55. Secondary Outcome: Extension Study: Percent Change From Baseline in the Affected BSA at Week 32
Description: as for outcome 16
Time Frame: Week 0 to Week 32
Population: Includes participants who entered the extension study and had a BSA assessment at Week 32; Intent to Treat
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 43 | 48 | 55 | 26 | 26
percent change | -47.1 (45.62) | -65.1 (30.42) | -75.3 (20.19) | -62.6 (29.48) | -66.7 (34.50)

56. Secondary Outcome: Extension Study: Percent Change From Baseline in the Affected BSA at Week 40
Description: as for outcome 16
Time Frame: Week 0 to Week 40
Population: Includes participants who entered the extension study and had BSA assessment at Week 40; Intent to Treat
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 36 | 40 | 51 | 24 | 21
percent change | -55.4 (33.33) | -65.4 (27.33) | -74.3 (17.98) | -66.2 (27.19) | -68.0 (32.83)

57. Secondary Outcome: Extension Study: Percent Change From Baseline in the Affected BSA at Week 52
Description: as for outcome 16
Time Frame: Week 0 to Week 52
Population: Includes participants who entered the extension study and had BSA assessment at Week 52; Intent to Treat;
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 34 | 34 | 49 | 22 | 19
percent change | -53.1 (30.33) | -58.3 (48.88) | -67.3 (32.56) | -67.4 (28.29) | -64.9 (31.26)

58. Secondary Outcome: Extension Study: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 32
Description: as for outcome 18
Time Frame: Week 0 to Week 32
Population: Includes participants who entered the extension study and had DLQI assessment at Week 32; Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 43 | 48 | 55 | 26 | 26
units on a scale | -6.5 (6.13) | -7.5 (6.20) | -6.0 (5.02) | -8.1 (7.16) | 5.5 (5.63)

59. Secondary Outcome: Extension Study: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 40
Description: as for outcome 18
Time Frame: Week 0 to Week 40
Population: Includes participants who entered the extension study and had DLQI assessment at Week 40; Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 36 | 40 | 52 | 23 | 21
units on a scale | -5.5 (6.42) | -6.6 (5.92) | -6.4 (4.51) | -7.1 (7.54) | -5.9 (5.03)

60. Secondary Outcome: Extension Study: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 52
Description: as for outcome 18
Time Frame: Week 0 to Week 52
Population: Includes participants who entered the extension study and had DLQI assessment at Week 40; Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 34 | 32 | 49 | 21 | 18
units on a scale | -5.8 (7.11) | -6.1 (5.14) | -5.6 (4.72) | -6.8 (7.16) | -4.9 (5.05)

61. Secondary Outcome: Extension Study: Change From Baseline in the Medical Outcome Study Short Form,SF-36, Version 2; Mental Component Summary Score at Week 32
Description: as for outcome 20
Time Frame: Week 0 to Week 32
Population: Includes participants who entered the extension study and had SF-36 assessment at Week 32; Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 43 | 48 | 54 | 25 | 26
units on a scale | 5.2 (9.45) | 3.8 (8.26) | 2.9 (7.80) | 4.6 (11.93) | 2.8 (9.64)

62. Secondary Outcome: Extension Study: Change From Baseline in the Medical Outcome Study Short Form,SF-36, Version 2; Physical Component Summary Score (PCS) at Week 32
Description: as for outcome 20
Time Frame: Week 0 to Week 32
Population: Includes participants who entered the extension study and had SF-36 assessment at Week 32; Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 43 | 48 | 54 | 25 | 26
units on a scale | 1.4 (5.26) | 2.6 (6.67) | 1.8 (7.58) | 3.1 (9.44) | 1.5 (8.46)

63. Secondary Outcome: Extension Study: Change From Baseline in the Medical Outcome Study Short Form,SF-36, Version 2; Mental Component Summary Score at Week 40
Description: as for outcome 20
Time Frame: Week 0 to Week 40
Population: Includes participants who entered the extension study and had SF-36 assessment at Week 40; Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 36 | 40 | 51 | 24 | 21
units on a scale | 5.4 (10.64) | 4.8 (8.95) | 1.7 (7.18) | 2.9 (12.24) | 3.8 (8.71)

64. Secondary Outcome: Extension Study: Change From Baseline in Medical Outcome Study Short Form,SF-36, Version 2; Physical Component Summary Score at Week 40
Description: as for outcome 20
Time Frame: Week 0 to Week 40
Population: Includes participants who entered the extension study and had SF-36 assessment at Week 40; Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 36 | 40 | 51 | 24 | 21
units on a scale | -0.2 (8.40) | 1.6 (7.77) | 1.7 (7.34) | 3.2 (10.89) | 1.8 (6.20)

65. Secondary Outcome: Extension Study: Change From Baseline in the Medical Outcome Study Short Form,SF-36, Version 2; Mental Component Summary Score at Week 52
Description: as for outcome 20
Time Frame: Week 0 to Week 52
Population: Includes participants who entered the extension study and had SF-36 assessment at Week 52; Intent to Treat;
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 34 | 33 | 49 | 21 | 19
units on a scale | 5.1 (11.56) | 4.1 (9.81) | 2.4 (7.91) | 4.7 (12.18) | 3.4 (7.49)

66. Secondary Outcome: Extension Study: Change From Baseline in the Medical Outcome Study Short Form,SF-36, Version 2; Physical Component Summary Score at Week 52
Description: as for outcome 20
Time Frame: Week 0 to Week 52
Population: Includes participants who entered the extension study and had SF-36 assessment at Week 52; Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 34 | 33 | 49 | 21 | 19
units on a scale | 1.2 (7.79) | 1.2 (5.50) | 2.0 (6.81) | 3.4 (12.84) | 0.3 (6.90)

67. Secondary Outcome: Extension Study: Dose-response Relationship Using the Percent Reduction of PASI Scores at Week 52
Description: Dose response relationship using percent reduction in PASI scores across dose groups at Week 52 compared to Week 0
Time Frame: Week 0 to Week 52
Population: The dose-response relationship analysis was anticipated, however, since the extension study was optional and there was not placebo control, no formal testing of dose response was conducted
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

68. Secondary Outcome: Extension Study: Time to Loss of Response During the Treatment Phase of the Extension Study.
Description: Time to 50% loss of the maximal improvement (achieved in either the core study or the extension study) during the treatment phase of the extension study, in participants who achieved ≥ PASI-50 in either the core study or during the treatment phase of the extension study
Time Frame: Week 0 to 52
Population: This endpoint was not summarized since the time of the maximal improvement is variable and the maximal improvement could occur in either the core phase or the extension phase
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

69. Secondary Outcome: Time to Loss of 50% of the PASI Response During the Observational Follow-up Phase Relative to the End of Treatment (Participants Who Had at Least a PASI-50 Response at the End of Treatment Phase)
Description: Time to loss of response was modified to be 50% loss in the PASI response observed at the end of treatment for participants who achieved at least a PASI-50 at the end of treatment. This definition was changed since participants may have already lost their maximal PASI response prior to enrollment into the Observation Follow-up Phase. Included all participants that enrolled into the observational follow-up phase after the treatment phase.
Time Frame: Up to 4 weeks after the last dose
Population: Participants who entered the observational follow-up phase and were PASI-50 responders at the beginning of the time interval.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 17 | 25 | 36 | 14 | 13
weeks | NA [4.3 to NA] — Not Available: the median and the limits of Confidence Interval (CI) could not be calculated due to insufficient number of participants who lost effect during the Observational Follow-up Phase. | NA [4.1 to NA] — Not Available: the median and the limits of Confidence Interval (CI) could not be calculated due to insufficient number of participants who lost effect during the Observational Follow-up Phase. | NA [4.3 to NA] — Not Available: the median and the limits of Confidence Interval (CI) could not be calculated due to insufficient number of participants who lost effect during the Observational Follow-up Phase. | NA [NA to NA] — Not Available: the median and the limits of Confidence Interval (CI) could not be calculated due to insufficient number of participants who lost effect during the Observational Follow-up Phase. | 5.3 [5.3 to NA] — Not Available: the median and the limits of Confidence Interval (CI) could not be calculated due to insufficient number of participants who lost effect during the Observational Follow-up Phase.

70. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) in the Placebo Controlled Phase
Description: An AE was any noxious, unintended, or untoward medical occurrence, that may appear or worsen in a participant during the course of study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) was considered an AE. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly/birth defect, or is a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above. An AE is a treatment emergent AE if the AE start date is on or after the date of the first dose of study drug and no later than 28 days after the last dose.
Time Frame: Week 0 to Week 16; up to data cut off of 21 July 2011
Population: Safety population consisted of all participants who were randomized and received at least one dose of Investigational Product (IP)
Measure: Number; unit: participants
Arm/Group | Placebo | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 88 | 89 | 87 | 88
participants
  Any treatment emergent AE | 57 | 59 | 67 | 72
  Any drug-related TEAE | 11 | 20 | 23 | 32
  Any severe TEAE | 3 | 1 | 5 | 5
  Any serious TEAE | 2 | 0 | 3 | 4
  Any serious drug-related | 0 | 0 | 0 | 0
  ≥ 1 TEAE leading to drug interruption | 4 | 3 | 3 | 6
  ≥ 1 TEAE leading to drug withdrawal | 5 | 2 | 8 | 12
  ≥ 1 TEAE leading to death | 1 | 0 | 0 | 0

71. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) in the Apremilast Exposure Period
Description: as for outcome 70
Time Frame: Week 0-88; up to data cut off of 21 July 2011
Population: Includes all participants who were treated with Apremilast
Measure: Number; unit: participants
Groups:
- Apremilast 10mg BID: Participants randomized to apremilast 10 mg PO BID during the Placebo-controlled Phase (Weeks 0-16) continued dosing with apremilast 10mg PO BID through Week 52 of the extension phase. Participants who received 10mg PO BID at the end of the extension study were randomly assigned to apremilast 20 mg or 30 mg PO BID during the long term extension study. (LTE).
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 89 | 121 | 124
participants
  Any treatment emergent AE | 67 | 97 | 110
  Any drug-related TEAE | 23 | 31 | 45
  Any severe TEAE | 3 | 9 | 13
  Any serious TEAE | 1 | 8 | 6
  Any serious drug-related | 0 | 1 | 0
  ≥ 1 TEAE leading to drug interruption | 3 | 11 | 9
  ≥ 1 TEAE leading to drug withdrawal | 5 | 11 | 15
  ≥ 1 TEAE leading to death | 0 | 0 | 0

72. Secondary Outcome: Core Study: Time to Achieve a PASI-50 Response During the Placebo Controlled Phase
Description: For PASI-50 responders in the placebo-controlled period weeks 0-16, time to achieve PASI-50 was defined as the time interval, inclusive between the date of randomization (day 1) and the date of the first assessment where PASI-50 was achieved.
Time Frame: Week 0 to 16
Population: Includes PASI-50 responders during the placebo controlled phase
Measure: Median (Full Range); unit: weeks
Groups:
- Placebo BID: Participants were initially randomized to placebo BID during the Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 28 | 49 | 49 | 59
weeks | 6.5 [2.1 to 16.9] | 5.9 [1.9 to 16.7] | 6.0 [2.1 to 16.4] | 4.3 [1.9 to 16.7]

73. Secondary Outcome: Core Study: Time to Achieve a PASI-75 Response During the Placebo Controlled Phase
Description: For PASI-75 responders in the placebo-controlled period Weeks 0-16, time to achieve PASI-75 was defined as the time interval, inclusive between the date of randomization (day 1) and the date of the first assessment where PASI-75 is achieved.
Time Frame: Weeks 0 to 16
Population: Includes PASI-75 responders during the placebo controlled phase.
Measure: Median (Full Range); unit: weeks
Groups:
- Placebo BID: .Participants were initially randomized to placebo PO BID during the Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 9 | 18 | 30 | 43
weeks | 8.1 [3.9 to 17.1] | 10.0 [4.0 to 16.0] | 11.9 [2.1 to 17.0] | 6.3 [3.7 to 16.7]

74. Secondary Outcome: Core Study: Time to Achieve a PASI-90 Response During the Placebo Controlled Phase
Description: For PASI-90 responders in the placebo-controlled period weeks 0-16, time to achieve PASI-90 was the time interval, inclusive, between the date of randomization (day 1) and the date of the first assessment where PASI-90 was achieved.
Time Frame: Weeks 0 to 16
Population: Time to achieve PASI-90 was not defined or analyzed as there were too few such participants.
Arm/Group | Placebo BID | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

75. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) in the Apremilast Exposure Period
Description: as for outcome 70
Time Frame: Week 0 to 6 years of study treatment; maximum duration of exposure was 314.6 weeks
Population: Safety population: includes all participants who were treated with Apremilast
Measure: Number; unit: participants
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 89 | 121 | 124
participants
  Any treatment emergent AE | 67 | 97 | 111
  Any drug-related TEAE | 23 | 32 | 46
  Any severe TEAE | 4 | 10 | 14
  Any serious TEAE | 2 | 9 | 6
  Any serious drug-related | 0 | 1 | 0
  ≥ 1 TEAE leading to drug interruption | 3 | 11 | 10
  ≥ 1 TEAE leading to drug withdrawal | 5 | 11 | 16
  ≥ 1 TEAE leading to death | 0 | 0 | 0

76. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 75% Improvement (Response) in the PASI Score at 18 Months
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Month 18
Population: ITT; participants who entered the long-term extension study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 60.0 [14.7 to 94.7] | 0.0 [0.0 to 60.2] | 40.0 [12.2 to 73.8] | 0.0 [0.0 to 60.2] | 50.0 [18.7 to 81.3]

77. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 75% Improvement (Response) in the PASI Score at 2 Years
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Month 24
Population: ITT; participants who entered the long-term extension study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 60.2] | 30.0 [6.7 to 65.2] | 25.0 [0.6 to 80.6] | 50.0 [18.7 to 81.3]

78. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 75% Improvement (Response) in the PASI Score at 3 Years
Description: as for outcome 76
Time Frame: Week 0 to Month 36
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 60.0 [14.7 to 94.7] | 25.0 [0.6 to 80.6] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 60.2] | 30.0 [6.7 to 65.2]

79. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 75% Improvement (Response) in the PASI Score at 4 Years
Description: as for outcome 76
Time Frame: Week 0 to Month 48
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 40.0 [5.3 to 85.3] | 0.0 [0.0 to 60.2] | 0 [0.0 to 30.8] | 25.0 [0.6 to 80.6] | 30.0 [6.7 to 65.2]

80. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score at 18 Months
Description: PASI-50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Month 18
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 100.0 [47.8 to 100.0] | 50.0 [6.8 to 93.2] | 70.0 [34.8 to 93.3] | 50.0 [6.8 to 93.2] | 100 [69.2 to 100.0]

81. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score at 2 Years
Description: as for outcome 80
Time Frame: Week 0 to Month 24
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 60.0 [14.7 to 94.7] | 50.0 [6.8 to 93.2] | 50.0 [18.7 to 81.3] | 25.0 [0.6 to 80.6] | 90.0 [55.5 to 99.7]

82. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score at 3 Years
Description: as for outcome 80
Time Frame: Week 0 to Month 36
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 60.0 [14.7 to 94.7] | 50.0 [6.8 to 93.2] | 30.0 [6.7 to 65.2] | 50.0 [6.8 to 93.2] | 60.0 [26.2 to 87.8]

83. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score at 4 Years
Description: as for outcome 80
Time Frame: Week 0 to Month 48
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 40.0 [5.3 to 85.3] | 25.0 [0.6 to 80.6] | 20.0 [2.5 to 55.6] | 25.0 [0.6 to 80.6] | 40.0 [12.2 to 73.8]

84. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 90% Improvement (Response) in the PASI Score at 18 Months
Description: PASI-90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 76 of the long-term extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Month 18
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 60.2] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 60.2] | 30.0 [6.7 to 65.2]

85. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 90% Improvement (Response) in the PASI Score at 2 Years
Description: PASI-90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 100 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Month 24
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 0.0 [0.0 to 52.2] | 0 [0.0 to 60.2] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 60.2] | 30.0 [6.7 to 65.2]

86. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 90% Improvement (Response) in the PASI Score at 3 Years
Description: PASI-90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 148 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Month 36
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 60.2] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 60.2] | 20.0 [2.5 to 55.6]

87. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 90% Improvement (Response) in the PASI Score at 4 Years
Description: PASI-90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 196 of the extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Month 48
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 60.2] | 20.0 [2.5 to 55.6]

88. Secondary Outcome: LTE Study: Percentage of Participants Who Achieved a 100% Improvement (Response) in the PASI Score at 18 Months, 2 Years, 3 Years and 4 Years
Description: PASI-100 response is the percentage of participants who achieved at a 100% reduction (improvement) from baseline in PASI score of the long-term extension study. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Week 0 to Month 48
Population: The PASI 100 was not defined and analyzed since there were too few such participants.
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

89. Secondary Outcome: LTE Study: Percent Change From Baseline in PASI Score at 18 Months
Description: as for outcome 11
Time Frame: Week 0 to Month 18
Population: ITT; Participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | PBO-Apremilast 20mg BID | Apremilast 20mg BID | PBO-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 2 | 10 | 4 | 10
percent change | -71.8 (14.84) | -60.5 (9.19) | -65.3 (21.28) | -50.0 (12.83) | -77.3 (17.77)

90. Secondary Outcome: LTE Study: Percent Change From Baseline in PASI Score at 2 Years
Description: as for outcome 11
Time Frame: Week 0 to Month 24
Population: ITT; Participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | PBO-Apremilast 20mg BID | Apremilast 20mg BID | PBO-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 2 | 7 | 4 | 9
percent change | -57.8 (19.51) | -64.5 (3.54) | -65.9 (21.22) | -46.0 (23.11) | -78.4 (16.60)

91. Secondary Outcome: LTE Study: Percent Change From Baseline in PASI Score at 3 Years
Description: as for outcome 11
Time Frame: Week 0 to Month 36
Population: ITT; Participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | PBO-Apremilast 20mg BID | Apremilast 20mg BID | PBO-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 3 | 2 | 6 | 4 | 6
percent change | -87.7 (5.69) | -69.0 (22.63) | -48.8 (29.69) | -48.0 (14.12) | -80.0 (17.88)

92. Secondary Outcome: LTE Study: Percent Change From Baseline in PASI Score at 4 Years
Description: as for outcome 11
Time Frame: Week 0 to Month 48
Population: ITT; Participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | PBO-Apremilast 20mg BID | Apremilast 20mg BID | PBO-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 4
percent change | -82.5 (0.71) | -52.0 (29.70) | -54.3 (20.55) | -80.0 (NA) — Standard Deviation is not available because there was only one participant analyzed. | -85.0 (17.80)

93. Secondary Outcome: Core Study: Shift Change (1 or More Points on a 0 to 5 Point Scale) in Static Physician Global Assessment (sPGA) at Month 18, and Years 2, 3 and 4
Description: as for outcome 14
Time Frame: Week 0 to Week 196
Population: as for outcome 15
Arm/Group | Apremilast 10mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 20 mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

94. Secondary Outcome: LTE Study: Percent Change From Baseline in the Percent of the Affected Body Surface Area (BSA) at 18 Months
Description: as for outcome 16
Time Frame: Week 0 to Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 2 | 10 | 4 | 10
percent change | -71.1 (16.82) | -73.9 (1.61) | -74.2 (18.83) | -44.2 (26.79) | -76.7 (23.70)

95. Secondary Outcome: LTE Study: Percent Change From Baseline in the Percent of the Affected Body Surface Area (BSA) at 2 Years
Description: as for outcome 16
Time Frame: Week 0 to Month 24
Population: ITT; participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 2 | 7 | 4 | 9
percent change | -64.7 (15.95) | -66.2 (3.62) | -74.5 (15.86) | -24.7 (49.99) | -74.5 (21.66)

96. Secondary Outcome: LTE Study: Percent Change From Baseline in the Percent of the Affected Body Surface Area (BSA) at 3 Years
Description: as for outcome 16
Time Frame: Week 0 to Month 36
Population: ITT; participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 3 | 2 | 6 | 4 | 6
percent change | -86.1 (3.00) | -63.4 (25.31) | -58.4 (29.80) | -39.1 (39.39) | -78.5 (21.02)

97. Secondary Outcome: LTE Study: Percent Change From Baseline in the Percent of the Affected Body Surface Area (BSA) at 4 Years
Description: as for outcome 16
Time Frame: Week 0 to Month 48
Population: ITT; participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 2 | 2 | 4 | 1 | 4
percent change | -75.0 (0.00) | -50.6 (18.48) | -72.4 (14.95) | -75.0 (NA) — Standard Deviation is not available because there was only one participant analyzed. | -86.1 (18.58)

98. Secondary Outcome: LTE Study: Median Percent Change From Baseline in the Affected Body Surface Area (BSA) at 18 Months
Description: as for outcome 16
Time Frame: Week 0 to Month 18
Population: Intent to Treat; participants who entered into the LTE period
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 2 | 10 | 4 | 10
percent change | -78.6 [-83.3 to -42.9] | -73.9 [-75.0 to -72.7] | -73.3 [-95.3 to -47.3] | -49.2 [-69.4 to -9.1] | -86.4 [-100.0 to -30.8]

99. Secondary Outcome: LTE Study: Median Percent Change From Baseline in the Affected Body Surface Area (BSA) at 2 Years
Description: as for outcome 16
Time Frame: Week 0 to Month 24
Population: Intent to Treat; participants who entered into the LTE period
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Apremilast 30 mg BID | Placebo-Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 2 | 7 | 4 | 9
percent change | -60.5 [-91.7 to -50.0] | -66.2 [-68.8 to -63.6] | -75.0 [-95.5 to -56.3] | -41.5 [-61.1 to 45.5] | -77.4 [-100.0 to -42.9]

100. Secondary Outcome: LTE Study: Median Percent Change From Baseline in the Affected Body Surface Area (BSA) at 3 Years
Description: as for outcome 16
Time Frame: Week 0 to Month 36
Population: Intent to Treat; participants who entered into the long-term extension period
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 3 | 2 | 6 | 4 | 6
percent change | -85.7 [-89.3 to -83.3] | -63.4 [-81.3 to -45.5] | -60.9 [-95.5 to -7.7] | -52.2 [-70.0 to 18.2] | -81.0 [-100.0 to -50.0]

101. Secondary Outcome: LTE Study: Median Percent Change From Baseline in the Affected Body Surface Area (BSA) at 4 Years
Description: as for outcome 16
Time Frame: Week 0 to Month 48
Population: Intent to Treat; participants who entered into the LTE period
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 2 | 2 | 4 | 1 | 4
percent change | -75.0 [-75.0 to -75.0] | -50.6 [-63.6 to -37.5] | -73.5 [-86.4 to -56.3] | -75.0 [-75.0 to -75.0] | -91.9 [-100.0 to -60.7]

102. Secondary Outcome: LTE Study: Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at 18 Months
Description: as for outcome 18
Time Frame: Week 0 to Month 18
Population: Intent to Treat; Includes participants who entered the long term extension period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
units on a scale |  |  | -6.5 (4.95) |  |

103. Secondary Outcome: LTE Study: Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at 2 Years
Description: as for outcome 18
Time Frame: Week 0 to Month 24
Population: Intent to Treat; Includes participants who entered the long term extension study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 2 | 7 | 4 | 9
units on a scale | -5.2 (5.17) | -13.5 (16.26) | -5.9 (5.70) | -1.8 (2.36) | -6.8 (4.27)

104. Secondary Outcome: LTE Study: Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at 3 Years
Description: as for outcome 18
Time Frame: Week 0 to Month 36
Population: Intent to Treat; Includes participants who entered the long term extension period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 3 | 1 | 6 | 4 | 6
units on a scale | -11.7 (5.03) | -3.0 (NA) — Standard Deviation is not available because there was only one participant analyzed. | -4.2 (3.37) | -2.0 (3.56) | -6.0 (6.03)

105. Secondary Outcome: LTE Study: Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at 4 Years
Description: as for outcome 18
Time Frame: Week 0 to Month 48
Population: Intent to Treat; Includes participants who entered the long term extension study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 2 | 2 | 4 | 1 | 3
units on a scale | -6.0 (5.66) | -9.0 (11.31) | -3.5 (1.00) | -7.0 (NA) — Standard Deviation is not available because there was only one participant analyzed. | -10.3 (5.13)

106. Secondary Outcome: LTE Study: Change From Baseline in the Medical Outcome Study Short Form, SF-36, Version 2; Mental Component Summary Score at 18 Months
Description: as for outcome 20
Time Frame: Week 0 to Month 18
Population: ITT; Includes participants who entered the long term extension period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
units on a scale |  |  | -2.8 (15.33) |  |

107. Secondary Outcome: LTE Study: Change From Baseline in the Medical Outcome Study Short Form, SF-36, Version 2; Mental Component Summary Score at 2 Years
Description: as for outcome 20
Time Frame: Week 0 to Month 24
Population: ITT; Includes participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 2 | 7 | 4 | 9
units on a scale | 5.0 (8.60) | 2.0 (14.75) | 5.2 (9.57) | 4.5 (8.75) | 0.2 (11.21)

108. Secondary Outcome: LTE Study: Change From Baseline in the Medical Outcome Study Short Form, SF-36, Version 2; Mental Component Summary Score at 3 Years
Description: as for outcome 20
Time Frame: Week 0 to Month 36
Population: ITT; Includes participants who entered the long-term extension study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 3 | 1 | 6 | 4 | 6
units on a scale | 6.0 (8.44) | -2.7 (NA) — Standard Deviation is not available because there was only one participant analyzed. | 3.6 (7.91) | 2.1 (10.79) | 2.4 (3.75)

109. Secondary Outcome: LTE Study: Change From Baseline in the Medical Outcome Study Short Form, SF-36, Version 2; Mental Component Summary Score at 4 Years
Description: as for outcome 20
Time Frame: Week 0 to Month 48
Population: ITT; Includes participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 2 | 2 | 4 | 1 | 4
units on a scale | -1.1 (19.83) | 4.1 (10.07) | -1.0 (1.50) | 17.6 (NA) — Standard Deviation is not available because there was only one participant analyzed. | 1.2 (6.54)

110. Secondary Outcome: LTE Study: Change From Baseline in the Medical Outcome Study Short Form,SF-36, Version 2; Physical Component Summary Score at 18 Months
Description: as for outcome 20
Time Frame: Week 0 to Month 18
Population: ITT; Includes participants who entered the long-term extension study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
units on a scale |  |  | 10.2 (11.84) |  |

111. Secondary Outcome: LTE Study: Change From Baseline in the Medical Outcome Study Short Form, SF-36, Version 2; Physical Component Summary Score at 2 Years
Description: as for outcome 20
Time Frame: Week 0 to Month 24
Population: ITT; Includes participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 2 | 7 | 4 | 9
units on a scale | 4.1 (9.15) | 3.7 (1.87) | 1.0 (7.13) | 2.4 (8.07) | 5.0 (6.33)

112. Secondary Outcome: LTE Study: Change From Baseline in the Medical Outcome Study Short Form, SF-36, Version 2; Physical Component Summary Score at 3 Years
Description: as for outcome 20
Time Frame: Week 0 to Month 36
Population: ITT; Includes participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 3 | 1 | 6 | 4 | 6
units on a scale | 6.6 (9.48) | 1.0 (NA) — Standard Deviation is not available because there was only one participant analyzed. | -0.1 (6.05) | 4.4 (7.49) | 4.2 (9.27)

113. Secondary Outcome: LTE Study: Change From Baseline in the Medical Outcome Study Short Form, SF-36, Version 2; Physical Component Summary Score at 4 Years
Description: as for outcome 20
Time Frame: Week 0 to Month 48
Population: ITT; Includes participants who entered the long-term extension period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 2 | 2 | 4 | 1 | 4
units on a scale | 1.4 (16.06) | 2.0 (0.79) | -4.1 (4.95) | 10.2 (NA) — Standard Deviation is not available because there was only one participant analyzed. | 9.4 (6.10)

114. Other Pre Specified Outcome: LTE Study: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of 0 or 1 at 18 Months
Description: as for outcome 12
Time Frame: Week 0 to Month 18
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 60.0 [14.7 to 94.7] | 0.0 [0.0 to 60.2] | 20.0 [2.5 to 55.6] | 25.0 [0.6 to 80.6] | 60.0 [26.2 to 87.8]

115. Other Pre Specified Outcome: LTE Study: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of 0 or 1 at 2 Years
Description: as for outcome 12
Time Frame: Week 0 to Month 24
Population: ITT; Participants who entered the extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 20.0 [0.5 to 71.6] | 0.00 [0.0 to 60.2] | 10.0 [0.3 to 44.5] | 25.0 [0.6 to 80.6] | 40.0 [12.2 to 73.8]

116. Other Pre Specified Outcome: LTE Study: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of 0 or 1 at 3 Years
Description: as for outcome 12
Time Frame: Week 0 and month 36
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 60.0 [14.7 to 94.7] | 0.0 [0.0 to 60.2] | 0 [0.0 to 30.8] | 25.0 [0.6 to 80.6] | 30.0 [6.7 to 65.2]

117. Other Pre Specified Outcome: LTE Study: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of 0 or 1 at 4 Years
Description: as for outcome 12
Time Frame: Week 0 to Month 48
Population: ITT; Participants who entered the long-term extension period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 10mg BID | Placebo-Apremilast 20 mg BID | Apremilast 20mg BID | Placebo-Apremilast 30 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 5 | 4 | 10 | 4 | 10
percentage of participants | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 30.8] | 25.0 [0.6 to 80.6] | 30.0 [6.7 to 65.2]

ADVERSE EVENTS:
Time Frame: Adverse Events are reported for the 16-week placebo-controlled phase and up to the LTE period, (6 years) for all participants who were randomized or re-randomized to apremilast at any time during the core, the extension or the long term extension study.
Description: Participants initially randomized to 10 mg PO BID were re-randomized at Week 52 to either 20 mg BID or 30 mg BID are included in the 10 mg BID group. Numbers of participants affected by serious adverse events were summarized. Some participants had more than one serious adverse event.
Groups:
- Placebo (Weeks 0-16): Participants randomized to placebo PO BID during the Placebo-controlled Phase
- Apremilast 10mg BID (Weeks 0-16): Participants randomized to apremilast 10 mg PO BID during the Placebo-controlled Phase (Weeks 0-16).
- Apremilast 20mg BID (Weeks 0-16): Participants randomized to apremilast 20 mg PO BID during the Placebo-controlled Phase (Weeks 0-16)
- Apremilast 30mg BID (Weeks 0-16): Participants randomized to apremilast 30 mg PO BID during the Placebo-controlled Phase (Weeks 0-16)
- Apremilast 10mg BID (APR Exposure Period) Years 0-6: Participants initially randomized to 10 mg PO BID apremilast at Week 0. Participants who were dosed with apremilast 10mg BID in the extension study were randomly assigned to either apremilast 20 mg or 30 mg BID in the long term extension study (LTE).
- Apremilast 20mg BID (APR Exposure Period) Years 0-6: Participants who received 20 mg PO BID apremilast, regardless of when the apremilast exposure started (at Week 0 or at Week 16 or Week 52), up to 6 years.
- Apremilast 30mg BID (APR Exposure Period) Years 0-6: Participants who received 30 mg PO BID apremilast, regardless of when the apremilast exposure started (at Week 0 or at Week 16 or Week 52), up to 6 years.
Arm/Group | Placebo (Weeks 0-16) | Apremilast 10mg BID (Weeks 0-16) | Apremilast 20mg BID (Weeks 0-16) | Apremilast 30mg BID (Weeks 0-16) | Apremilast 10mg BID (APR Exposure Period) Years 0-6 | Apremilast 20mg BID (APR Exposure Period) Years 0-6 | Apremilast 30mg BID (APR Exposure Period) Years 0-6
Serious Adverse Events (participants affected / at risk) | 2/88 | 0/89 | 3/87 | 4/88 | 2/89 | 9/121 | 9/124
Other Adverse Events (participants affected / at risk) | 35/88 | 42/89 | 45/87 | 55/88 | 52/89 | 66/121 | 85/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-16) (N=88) | Apremilast 10mg BID (Weeks 0-16) (N=89) | Apremilast 20mg BID (Weeks 0-16) (N=87) | Apremilast 30mg BID (Weeks 0-16) (N=88) | Apremilast 10mg BID (APR Exposure Period) Years 0-6 (N=89) | Apremilast 20mg BID (APR Exposure Period) Years 0-6 (N=121) | Apremilast 30mg BID (APR Exposure Period) Years 0-6 (N=124)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-16) (N=88) | Apremilast 10mg BID (Weeks 0-16) (N=89) | Apremilast 20mg BID (Weeks 0-16) (N=87) | Apremilast 30mg BID (Weeks 0-16) (N=88) | Apremilast 10mg BID (APR Exposure Period) Years 0-6 (N=89) | Apremilast 20mg BID (APR Exposure Period) Years 0-6 (N=121) | Apremilast 30mg BID (APR Exposure Period) Years 0-6 (N=124)
Diarrhoea (Gastrointestinal disorders) | 4 | 6 | 6 | 12 | 7 | 9 | 17
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 5 | 4 | 1 | 6 | 9
Nausea (Gastrointestinal disorders) | 7 | 10 | 13 | 17 | 12 | 20 | 28
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 4 | 1 | 8 | 5
Gastroenteritis (Infections and infestations) | 3 | 1 | 4 | 5 | 4 | 8 | 7
Nasopharyngitis (Infections and infestations) | 7 | 8 | 7 | 5 | 10 | 11 | 13
Sinusitis (Infections and infestations) | 2 | 3 | 0 | 3 | 5 | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 4 | 9 | 11 | 14 | 14 | 19 | 25
Viral upper respiratory tract infection (Infections and infestations) | 8 | 2 | 8 | 7 | 7 | 13 | 13
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0 | 5 | 5 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0 | 1 | 0 | 2 | 1
Headache (Nervous system disorders) | 5 | 5 | 8 | 7 | 7 | 13 | 11
Tension headache (Nervous system disorders) | 7 | 3 | 2 | 14 | 4 | 4 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.